CLINICAL TRIAL: NCT04789018
Title: Enhanced Genetic Awareness and Genetic Evaluation for Men Through Technology ENGAGEMENT Study (Virtual Genetics Board)
Brief Title: Enhanced Genetic Awareness and Genetic Evaluation for Men Through Technology, ENGAGEMENT Study
Status: Active, not recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 20F.936; JT 16041 (Other: JeffTrial Number); 080-27000-X17501 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2021-02-19; First posted 2021-03-09 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey, virtual genetic board, interview): Participants complete a survey about genetic knowledge and self efficacy and then attend virtual genetics board. After virtual genetics board meeting, participants complete a second survey about perceived usefulness, ease of use, acceptability, feasibility, self-efficacy and genetic knowledge. Participants may also complete a semi-structured interview after virtual genetics board.
  Interventions: Other: Educational Intervention; Other: Survey Administration; Other: Interview

INTERVENTIONS:
Other: Educational Intervention — Attend virtual genetics board
  Other Names: Education for Intervention, Intervention by Education, Intervention through Education, Intervention, Educational
Other: Survey Administration — Complete survey
Other: Interview — Complete interview

SUMMARY:
This study assesses perceived usefulness of a web-based virtual prostate cancer genetics board for providers across academic, community, and veteran affairs settings to discuss prostate cancer genetics cases, precision treatment, and screening recommendation. Information gained from interviews and surveys of participants taking part in the virtual genetics board may lend insights into perceived usefulness, perceived ease of use, acceptability, self-efficacy, genetics knowledge, and barriers/facilitators to implementation to refine the process.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess perceived usefulness of a virtual genetics board.

SECONDARY OBJECTIVE:

I. To assess acceptability/feasibility, perceived ease of use, self-efficacy for recommendations, genetics knowledge.

OUTLINE:

Participants complete a survey about genetic knowledge and self efficacy and then attend virtual genetics board. After virtual genetics board meeting, participants complete a second survey about perceived usefulness, ease of use, acceptability, feasibility, self-efficacy and genetic knowledge. Participants may also complete a semi-structured interview after virtual genetics board.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet one of the following inclusion criteria in order to be eligible to participate in the study:

* Healthcare providers (medical oncologists, radiation oncologists, urologists, primary care providers, mid-level providers) who evaluate, manage, or treat men with prostate cancer or screen men for prostate cancer.
* Providers who perform prostate cancer genetic testing for men (genetic counselors or healthcare providers)
* Scientists and researchers
* Advocacy or patient stakeholder organization members

Exclusion Criteria:

• Non-medical providers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-genetic providers who perform prostate cancer (PCA) genetic testing for men in their practices (medical oncologists, radiation oncologists, urologists, primary care providers, mid-level providers)
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Mean Likert scaled perceived usefulness scores of the virtual genetics board | After virtual genetics board
  Perceived usefulness will be judged against a benchmark mean score of 5/7.

SECONDARY OUTCOMES:
Means or changes in means of Likert scaled acceptability/feasibility | Before and after virtual genetics board
  Will be summarized by means, standard deviations, and 95% confidence intervals.
Perceived ease of use | After virtual genetics board
  Will be summarized by means, standard deviations, and 95% confidence intervals.
Self-efficacy for recommendations | Before and after virtual genetics board
  Will be summarized by means, standard deviations, and 95% confidence intervals.
Change in mean scores on 17 genetics knowledge test questions | Baseline up to post-virtual genetics board
  Will be summarized by means, standard deviations, and 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Leader, DrPH, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No